CLINICAL TRIAL: NCT06050694
Title: Feasibility Trial of Glofitamab in a Response Adapted Approach Incorporating Interim FDG PET and ctDNA to Optimize Primary Therapy of DLBCL
Brief Title: Feasibility Trial of Glofitamab in a Response Adapted Approach Incorporating Interim FDG PET and ctDNA to Optimize Primary Therapy of DLBCL (GRAIL)
Acronym: GRAIL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: OZM-121
Record Dates: First submitted 2023-08-29; First posted 2023-09-22 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — glofitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pola-R-CHP (No Intervention): Protocol induction: Cycle 1-2
  Low-risk group: Cycle 3-4 polatuzumab vedotin 1.8 mg/kg, cyclophosphamide 750 mg/m2 and doxorubicin 50 mg/m2 on day 1, prednisone 100 mg daily days 1-5, and rituximab 375 mg/m2 within 72 hours of polatuzumab vedotin
  Cycle 5-6 rituximab 375 mg/m2 on day 1 of cycle 5 and cycle 6
- Pola-R-CHP and glofitamab (Experimental): High-risk group: Cycle 3-6 polatuzumab vedotin 1.8 mg/kg, cyclophosphamide 750 mg/m2 and doxorubicin 50 mg/m2 on day 1, prednisone 100 mg daily days 1-5, rituximab 375 mg/m2 within 72 hours of polatuzumab vedotin and Glofitamab 2.5 mg Cycle 3 Day 8 and 10 mg on Day 15 Cycles 3-6
  Interventions: Drug: glofitamab

INTERVENTIONS:
Drug: glofitamab — Glofitamab 2.5 mg Cycle 3 Day 8 and 10 mg on Day 15 Cycles 3-6
  Arms: Pola-R-CHP and glofitamab

SUMMARY:
This is a phase ll study of participants with untreated diffuse large B Cell lymphoma (DLBCL).

DETAILED DESCRIPTION:
This is a multicenter, phase II, non-randomized, open-label, single-arm study in patients with untreated DLBCL. Patients will be on treatment for a total of 6 cycles, each 21 days in length.

After receiving 2 cycles of polatuzumab vedotin, cyclophosphamide, doxorubicin, prednisone (Pola-R-CHP), a risk-adapted approach will be used to modify therapy for patients who are found to be of an unfavourable risk. Pola-R-CHP chemotherapy will be administered every 21 days at standard doses: polatuzumab vedotin 1.8 mg/kg IV on day 1, cyclophosphamide 750 mg/m2 IV on day 1, doxorubicin 50 mg/m2 IV on day 1, prednisone 100 mg orally daily days 1-5, and rituximab 375 mg/m2 IV within 72 hours of polatuzumab vedotin and CHP. No subcutaneous administration of rituximab is allowed in this study.

All patients will undergo circulating tumour DNA (ctDNA) evaluation in peripheral blood at baseline and prior to cycle 2 of Pola-R-CHP. Interim response will also be assessed by 18-fluorodeoxyglucose positron emission tomography (FDG-PET) scan response prior to cycle 3 of treatment positron emission tomography (PET2). Based on these tests, patients will be risk stratified into two treatment arms. The ctDNA low-risk patients (favourable ctDNA and PET2) will receive two additional cycles of Pola-R-CHP chemotherapy followed by 2 additional courses of rituximab. See Table 3 for exact treatment dosing for Cycles 3 - 6.

The ctDNA high-risk risk group (unfavourable ctDNA and/or PET2) will receive 4 additional cycles of Pola-R-CHP chemotherapy given with glofitamab. See Table 4 for exact treatment dosing for Cycles 3 - 6. Following six cycles of treatment, patients in both groups will undergo treatment assessment with CT scan, PET/CT scan, and bone marrow biopsy (as required).

Following completion of protocol treatment, patients will go into survival follow-up. Routine assessments will include patient visits with laboratory testing including ctDNA testing every 3 months. Imaging studies (PET/CT scan) will be repeated every 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age deemed eligible for treatment with full-dose Pola- R-CHP and possible treatment with glofitamab by the qualified investigator.
2. Histologic diagnosis of DLBCL and variants according to the WHO 201613 or WHO 202254 classification including DLBCL non-organ-specific (NOS), Germinal centre B-cell type, activated B-cell type, T-cell/histiocyte-rich large B-cell lymphoma, Epstein-Barr Virus (EBV) + DLBCL, Primary mediastinal/thymic large B-cell lymphoma, High grade B-cell lymphoma with myelocytomatosis oncogene (MYC) and B-cell lymphoma 2 (BCL2) and/or B-cell lymphoma 6 (BCL6) rearrangements, High grade B cell lymphoma NOS including lymphomas transformed from previously untreated indolent lymphomas.
3. Previously untreated DLBCL with the following exceptions: (a) prior radiotherapy for palliation (not localized), (b) up to 7 days of corticosteroids (prednisone 100mg/day equivalent).
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
5. Presence of at least one radiologically measurable nodal or extranodal mass. A measurable nodal mass must have a longest diameter ≥1.5 cm. A measurable extranodal mass should have a longest diameter ≥1.0 cm.16
6. Left ventricular ejection fraction (LVEF) ≥ 50%, as determined on cardiac multiple- gated acquisition (MUGA) scan or cardiac echocardiogram (ECHO)
7. Women of childbearing potential (WOCBP) who are sexually active must use highly effective methods of contraception during treatment and up to 18 months after the last dose of or protocol therapy. Men who are sexually active must use highly effective methods of contraception during treatment and up to 6 months after the last dose of protocol therapy. Men require an agreement to remain abstinent (ie, refrain from heterosexual intercourse) or use a condom, and an agreement to refrain from donating sperm. Periodic abstinence and withdrawal are not acceptable methods of contraception. Fertility preservation options should be discussed. Examples of highly effective contraceptive methods include an agreement to remain abstinent (ie, refrain from heterosexual intercourse), bilateral tubal ligation, male sterilization, established proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
8. Willing and able to participate in all required evaluations and procedures in this study.
9. Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained by the patient or legally acceptable representative before any study-specific procedures are performed.

Exclusion Criteria:

1. Current/past history of central nervous system (CNS) lymphoma.
2. Prior exposure to any anthracycline, rituximab or cluster of differentiation 3 (CD3) targeted bispecific antibody.
3. Prior malignancy (or any other malignancy requiring active treatment), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease free for ≥ 2 years or which will not limit survival to < 5 years. Subjects receiving adjuvant hormonal therapy for early breast or prostate cancer are eligible.
4. Significant or extensive cardiovascular disease such as New York Heart Association Class III or IV cardiac disease or Objective Assessment Class C or D, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina. Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll on study.
5. Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including diabetes mellitus, history of relevant pulmonary disorders (bronchospasm, obstructive pulmonary disease), and known autoimmune diseases.
6. Patients with a known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
7. History of illicit drug or alcohol abuse within 12 months prior to screening, in the Investigator's judgment.
8. Known active infection, or reactivation of a latent infection, whether bacterial, viral (including, but not limited to, EBV, cytomegalovirus (CMV), hepatitis B, hepatitis C, and human immunodeficiency virus (HIV), fungal, mycobacterial, or other pathogens (excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics (for IV antibiotics this pertains to completion of last course of antibiotic treatment) within 4 weeks of dosing. Individuals with a positive HIV test at screening are eligible provided they are stable on antiretroviral therapy, have a cluster of differentiation 4 (CD4) count ≥ 200/μL, and have an undetectable viral load. HIV positive patients should be monitored per local/institutional standards while receiving study treatment.
9. Known history of drug-specific hypersensitivity or anaphylaxis to study drugs (glofitamab and individual components of Pola-R-CHP), including grade III or greater allergic reactions to any monoclonal antibody.
10. Known Type I hypersensitivity or anaphylactic reactions to murine proteins, Chinese Hamster Ovary (CHO) cell proteins, or to any component of Rituximab
11. Current history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease. Patients with a history of stroke who have not experienced a stroke or transient ischemic attack within the past 2 years and have no residual neurological deficient, as judged by the investigator, are allowed.
12. Active autoimmune disease which is not well controlled by therapy:

    * Participants with a history of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone may be eligible. Participants with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
    * Participants with active autoimmune disease with dermatologic manifestations are eligible for the study.
    * Participants with a history of autoimmune hepatitis, systemic lupus erythematosus, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener granulomatosis, Sjögren syndrome, multiple sclerosis, or glomerulonephritis will be excluded.
    * Participants with a history of immune thrombocytopenic purpura, autoimmune hemolytic anemia, Guillain-Barré syndrome, myasthenia gravis, myositis, rheumatoid arthritis, vasculitis, or other autoimmune disease will be excluded unless they have not required systemic therapy in the last 12 months
13. Major surgical procedure within 4 weeks of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
14. Administration of a live, attenuated vaccine within 4 weeks before study treatment infusion on Cycle 1/Day 1 or anticipation that such a live, attenuated vaccine will be required during the study. Live vaccines during the study and until participants' B- cells recover, are prohibited. Note: Influenza vaccination should be given during influenza season only. Participants must not receive live, attenuated influenza vaccine (e.g., FluMist) at any time during the study treatment period).
15. Use of any of the prohibited therapies including: investigational or unlicensed/unapproved agents; biologic agents (e.g., bevacizumab, erlotinib); immunotherapy/radio-immunotherapy; radiotherapy (with the exception of limited field palliative radiotherapy for bone pain or for soft tissue lesions after consultation with the Sponsor); chemotherapy (apart from Pola-R-CHP per protocol); hormone therapy (other than contraceptives, hormone-replacement therapy, or megestrol acetate); chronic use of steroids (inhaled, topical or systemic)
16. Positive test results for hepatitis B virus (HBV) infection (defined as positive B surface antigen [HBsAg] serology). Patients with occult or prior HBV infection (defined as negative HBsAg and positive hepatitis B core antibody [HBcAb]) may be included if HBV DNA is undetectable, provided that they are willing to undergo DNA testing on Day 1 of every cycle and every three months for at least 12 months after the last cycle of study treatment and appropriate antiviral therapy.
17. Positive test results for hepatitis C virus (HCV) antibody. Patients who are positive for HCV antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.
18. Absolute Neutrophil Count (ANC) <1.0 x109/L (subjects with bone marrow involvement by lymphoma are eligible regardless of ANC).
19. Hemoglobin (Hgb) ≤ 9 g/dL
20. Platelets <50 x109/L (subjects with bone marrow involvement by lymphoma are eligible regardless of platelet count)
21. Total serum bilirubin >2 times the upper limit of normal (or <3 times for Gilbert's disease or documented hepatic involvement by lymphoma), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >3 times the upper limit of normal (or >5 times for documented hepatic involvement by lymphoma)
22. Creatinine clearance <30 mL/min.
23. Prothrombin time (PT)/ international normalized ratio (INR) >2 times the upper limit of normal in the absence of anticoagulants or partial thromboplastin time (PTT) >2 times the upper limit of normal in the absence of anticoagulants.
24. Breastfeeding or pregnant, or intending to become pregnant during the study or within 12 months after the final dose of Pola-R-CHP, 3 months after the final dose of tocilizumab (if applicable), or 2 months after the final dose of glofitamab. WOCBP must have a serum pregnancy test done a maximum of 7 days prior to treatment initiation and a negative result must be documented prior to recruitment.
25. Concurrent participation in another therapeutic clinical trial.
26. Any other diseases, metabolic dysfunction, physical examination finding, or clinical
27. Laboratory finding giving reasonable suspicion of a disease or condition that would contraindicate the use of an investigational drug.
28. Current Grade > 1 peripheral neuropathy by clinical examination or demyelinating form of Charcot Marie Tooth disease.
29. Known history of progressive multifocal leukoencephalopathy.
30. Positive severe acute respiratory syndrome (SARS-CoV-2) test within 7 days prior to enrollment. Rapid antigen test result is also acceptable.
31. Known or suspected chronic active Epstein-Barr viral infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the feasibility of a ctDNA and FDG-PET interim response adapted approach (iRAAp) for the primary therapy of DLBCL | At the end of cycle 1 (ctDNA) and cycle 2 (PET)(each cycle is 21 days)
  Determine the proportion of patients that can have results available to risk adapt cycle treatment starting at cycle 3 based on interim testing (ctDNA collected immediately prior to cycle 2 of Pola-R-CHP, PET scan following cycle 2 of Pola-R-CHP ie. PET2). Treat the ctDNA low-risk patients (favourable ctDNA and PET2) with abbreviated chemotherapy (total 4 cycles of Pola-R-CHP with 2 courses of rituximab as a monotherapy). Treat the ctDNA high-risk patients (unfavourable ctDNA and/or PET2) with a novel treatment approach (complete 3 cycles of Pola-R-CHP and then start novel approach).

SECONDARY OUTCOMES:
Event-free survival (EFS) | baseline to month 24
  To evaluate the event-free survival (EFS) of an iRAAp in primary therapy of DLBCL
Incidence of treatment emergent adverse events | baseline to cycle 6 (each cycle is 21 days)
  To evaluate the tolerability and toxicity of an iRAAp in primary therapy of DLBCL by assessing the frequency, severity, and relatedness of adverse events
Progression free survival (PFS) at 12 months and 24 months | baseline to 24 months
  To assess PFS at 12-months and 24-months in the whole population and both ctDNA high-risk and ctDNA low-risk response cohorts.
To evaluate changes in health-related quality of life (HRQOL) | baseline through year 2
  To evaluate changes in health-related quality of life (HRQOL) through treatment and follow-up. HRQOL inclusive of three validated patient-reported outcome (PRO) instruments (FACT-Lym, FACT-Cog and EORTC QLQ-C30) that will be completed by the participant at required visits. The FACT-Lym was designed to address health-related quality-of-life issues for patients with non-Hodgkin's lymphoma (NHL), and includes both general concerns related to cancer treatments and specific concerns relevant to lymphoma. The FACT-Cog is a well-validated tool that measures cognitive complaints. The EORTC QLQ-C30 includes 30 separate questions (items) resulting in 5 functional scales (Physical Functioning, Role Functioning, Emotional Functioning, Cognitive Functioning, and Social Functioning), 1 Global Health Status scale, 3 symptom scales (Fatigue, Nausea and Vomiting, and Pain), and 6 single items (Dyspnea, Insomnia, Appetite Loss, Constipation, Diarrhea, and Financial Difficulties).
Overall survival (OS) at 12 months and 24 months | baseline to 24 months
  To assess OS at 12-months and 24 months in the whole population and both ctDNA high-risk and ctDNA low-risk response cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: John Kuruvilla, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No